CLINICAL TRIAL: NCT02865473
Title: Anterior Segment Imaging With Ultrahigh-resolution OCT in Patients With Glaucoma and Pseudoexfoliation Syndrome - a Pilot Study
Brief Title: Anterior Segment Imaging With Ultrahigh-resolution OCT in Patients With Glaucoma and PEX - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-010915
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma
Keywords: Schlemm's canal lumen area; PEX
MeSH Terms: conditions — Glaucoma | interventions — Pilocarpine

ARMS (6):
- primary open angle glaucoma patients (No Intervention)
- patients with primary angle closure (No Intervention)
- patients with neovascular glaucoma (No Intervention)
- PEX glaucoma patients (No Intervention)
- glaucoma patients with filtering bleb (No Intervention)
- healthy volunteers (Experimental): instillation of antiglaucoma treatment in the study eye
  Interventions: Drug: Pilocarpine

INTERVENTIONS:
Drug: Pilocarpine — topical instillation into the study eye
  Arms: healthy volunteers

SUMMARY:
The aim of the present study is to develop a measurement protocol for optimal imaging of the anterior segment of the eye, including anterior chamber angle, Schlemm's canal, filtering bleb and pseudoexfoliation deposits on the lens based on measurements in patients with glaucoma and PEX. In glaucoma the structures of the anterior chamber are important for classification, therapy, progression and prognosis and imaging of the angle between the iris and the cornea is the key for open angle and closed angle glaucoma differential diagnosis. For this purpose, a customized ultrahigh resolution Spectral Domain OCT will be used to validate whether the protocol can also be more widely applied in these patients. Based on the obtained measurement protocol, further studies investigating anatomy and pathophysiology of the anterior segment of the eye as well as surgical outcome in patients with glaucoma and PEX can be planned.

The aim of the study is to develop a measurement protocol for OCT imaging and characterization of the anterior chamber in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years

For patients with primary open angle glaucoma:

* Diagnosed primary open angle glaucoma
* Visual field defects and optic nerve head appearance characteristic for glaucoma
* Open anterior chamber angle as evidenced by gonioscopy
* No previous glaucoma surgery
* No previous cataract surgery

For patients with primary angle closure:

* Angle closure predisposition as evidenced from goniosocopy
* No previous glaucoma surgery

For patients with neovascular glaucoma:

- Neovascularization in the anterior chamber angle

For patients with pseudoexfolation deposits on the lens:

* PEX glaucoma as evidenced from slit lamp examination
* Visual field defects and optic nerve head appearance characteristic for glaucoma
* Open anterior chamber angle as evidenced by gonioscopy
* No previous glaucoma or cataract surgery

For glaucoma patients with filtering bleb after trabeculectomy:

* Patients with history of trabeculectomy secondary to open angle glaucoma in the previous three months
* No cataract surgery

For healthy volunteers:

* No evidence of ocular disease
* No degenerative changes in the retina in funduscopy after mydriasis
* Ametropia less than 3 dpt.

Exclusion Criteria:

* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating
* Ocular inflammation and ocular disease interfering with the study aims as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-04-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3-dimensional imaging of the anterior eye segment | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria